CLINICAL TRIAL: NCT06244134
Title: Ultrasound -Guided Versus Conventional Non Guided Autologous Blood Injection For Treatment of Patients With Chronic Recurrent Temporomandibular Joint Dislocation. A Randomized Clinical Trial
Brief Title: Ultrasound Guided Autologous Blood Injection in Temporomandibular Joint Dislocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abbas Morsy Hussien, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 291123
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Temporomandibular Joint Dislocation
Keywords: ultrasound; autologous blood; temporomandibular joint; dislocation
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (group A) will be injected with ultrasound guidance in temporomandibular joint . (Active Comparator): uses of ultrasound as a guiding tool for temporomandibular joint injection
  Interventions: Procedure: ultrasound guided autologous blood injection
- control group(group B) conventional non guided injection in temporomandibular joint (Placebo Comparator): without ultrasound guidance only anatomical landmark will be followed during injection
  Interventions: Procedure: non guided autologous blood injection

INTERVENTIONS:
Procedure: ultrasound guided autologous blood injection — guided
  Arms: Study group (group A) will be injected with ultrasound guidance in temporomandibular joint .
Procedure: non guided autologous blood injection — non guided
  Arms: control group(group B) conventional non guided injection in temporomandibular joint

SUMMARY:
The aim of this study is To compare the accuracy and effectiveness of ultrasound (US) guided autologous blood injection (ABI) versus non- guided technique for the treatment of chronic recurrent temporomandibular joint dislocation

DETAILED DESCRIPTION:
All patients involved in this study will be divided randomly to two different groups and injected with autologous blood into joint space and pericapsular tissue.

Study group (group A) will be injected with autologous blood with ultrasound guidance.

control group (group B) will be injected with autologous blood without US guidance. Anatomical landmarks and tactical sense will be followed only.

The operation will be done under local anesthesia ( Auriculotemporal nerve block ) the skin overlying the temporomandibular joint will be scrubbed by an antiseptic solution and the area will be isolated with sterile towels. External auditory canal will be blocked with cotton.

About 3 ml of blood will be withdrawn from patient's antecubital fossa, of which 2 ml injected intra-articular and 1 ml in the pericapsular tissue (PT) The procedure should be repeated on the opposite side in case of bilateral involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient with at least 3 episodes of temporomandibular joint dislocation in the past 6 months.
* Necessitating a visit to the emergency room or trained professional to reduce the dislocation.
* Radiological evidence of displacement of condylar head beyond the articular eminence on wide mouth opening.
* Maximum mouth opening (MMO) more than 40 mm.
* Unilateral or bilateral.
* Over 18 years of age.
* Both gender Males or females.

Exclusion Criteria:

* Patient having inflammatory temporomandibular joint disease like tuberculous arthritis, rheumatoid arthritis.
* Patients with bleeding disorders, pregnancy or bony pathology of temporomandibular joint .
* Allergy to local anesthetic.
* Severe epilepsy or Parkinson's disease.
* Patient on anti-depressants or anti-psychotics.
* Inability to follow-up the patient during the entire follow-up period.
* Patients who had recent fracture at temporomandibular joint level or who had previous surgical interference to temporomandibular joint .
* Refused to sign the written informed consent were also excluded.
* Dystonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
maximum mouth opening | at 2weeks, 3months and 6 months post-operative
  change in Maximum mouth opening (MMO): It's measured (in millimeter) from incisal edge of 11 to 41, in maximum mouth open position using caliper

SECONDARY OUTCOMES:
Frequency of temporomandibular joint dislocation: | 2weeks, 3 months and 6 months post-operatively
  number of dislocation per week
change of pain | 2weeks, 3 months and 6 months post-operatively
  measuring pain using visual analogue scale(0-10),higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Gagnani SP, Kholakiya YR, Arora A, Bhutia O, Seith A, Khandelwal RK, Roychoudhury A. Ultrasound-guided autologous blood injection in patients with chronic recurrent temporomandibular joint dislocation. Natl J Maxillofac Surg. 2020 Jan-Jun;11(1):34-39. doi: 10.4103/njms.NJMS_57_18. Epub 2020 Jun 18. PMID 33041574
- [Background] Pandey SK, Baidya M, Srivastava A, Garg H. Comparison of autologous blood prolotherapy and 25% dextrose prolotherapy for the treatment of chronic recurrent temporomandibular joint dislocation on the basis of clinical parameters: A retrospective study. Natl J Maxillofac Surg. 2022 Sep-Dec;13(3):398-404. doi: 10.4103/njms.njms_509_21. Epub 2022 Dec 10. PMID 36683930